CLINICAL TRIAL: NCT02579616
Title: An Open-Label, Multicenter Phase 2 Study of E7080/ LENVIMA (Lenvatinib Mesylate) in Subjects With Unresectable Biliary Tract Cancer Who Failed Gemcitabine-based Combination Chemotherapy
Brief Title: Study of Lenvatinib (E7080) in Unresectable Biliary Tract Cancer (BTC) Who Failed Gemcitabine-based Combination Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-215
Record Dates: First submitted 2015-10-16; First posted 2015-10-19 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-10

CONDITIONS: Biliary Tract Cancer
Keywords: Lenvatinib; E7080; Unresectable biliary tract cancer; BTC; Gemcitabine-based combination chemotherapy; Lenvima
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 24 mg Lenvatinib (Experimental): Participants with unresectable BTC and disease progression or failure following one prior gemcitabine-based doublet chemotherapy regimen (combination of gemcitabine and cisplatin, or gemcitabine and other platinum agent/fluoropyrimidine agent).
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be administered orally once daily in 28-day cycles. Participants will be treated until disease progression, unacceptable toxicity, withdrawal of consent, participant's choice, etc.
  Other Names: E7080; Lenvima; Lenvatinib Mesylate

SUMMARY:
This is a multicenter, single arm, open-label study in participants with unresectable BTC and disease progression or failure following one prior gemcitabine-based doublet chemotherapy regimen (combination of gemcitabine and cisplatin, or gemcitabine and other platinum agent/fluoropyrimidine agent). This study contains 3 phases: a Pre-treatment phase that will last within 21 days; a Treatment phase that will consist of study treatment cycles and tumor assessment conducted every 6-8 weeks; and a Follow-up phase that will begin immediately after the Off-Treatment Visit and will continue as long as the participant is alive, unless the participant withdraws consent, or until the End of Study.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed adenocarcinoma of biliary tract cancer (intrahepatic, extrahepatic cholangiocarcinoma, gall bladder cancer, and ampulla of Vater cancer)
2. Unresectable (eg, locally advanced or metastatic) BTC
3. One prior gemcitabine-based doublet chemotherapy (eg, gemcitabine and cisplatin) to unresectable BTC and not treated by any other chemotherapy to BTC

   * Participants who received adjuvant chemotherapy are eligible if this therapy was completed and recurrent has not been shown for 6 months after the completion of the therapy
4. Measurable disease meeting the following criteria:

   * At least 1 lesion of ≥ 1.0 cm in the longest diameter for a non-lymph node or ≥ 1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST1.1) using computerized tomography/magnetic resonance imaging (CT/MRI)
   * Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
6. Survival expectation of 3 months or longer after beginning of study treatment
7. Males or females age ≥ 20 years at the time of informed consent
8. All chemotherapy- or radiation-related toxicities must have resolved to Grade 0-1 per Common Terminology Criteria for Adverse Events (CTCAE v 4.03), except alopecia, infertility, and the adverse events listed in inclusion criteria
9. Adequately controlled blood pressure (BP) with or without antihypertensive medications (defined as BP ≤ 150/90 mm Hg at Screening and no change in antihypertensive medications within 1 week prior to the first dose of study drug)
10. Participants with adequate function of major organs and blood coagulation:

    * Absolute neutrophil count (ANC) ≥ 1500/mm^3 ( ≥ 1.5×103/μl)
    * Platelets ≥ 100,000/mm3 ( ≥ 100×10^9/L)
    * Hemoglobin ≥ 9.0 g/dL
    * Bilirubin ≤ 2.0 mg/dL except for unconjugated hyperbilirubinemia or Gilbert's syndrome
    * Alkaline phosphatase (ALP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN) ( ≤ 5.0 × ULN for participants with the liver metastasis)
    * Creatinine clearance ≥ 40 mL/min per the Cockcroft and Gault formula
    * Prothrombin time-International Normalized Ratio (PT-INR) ≤ 1.5
11. Participants must voluntarily agree to provide written informed consent
12. Participants must be willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Any anti-cancer treatment (except BSC) within 21 days prior to the first dose of study drug
2. Major surgery (any surgical procedure that involves anesthesia or respiratory assistance) within 21 days prior to the first dose of study drug or scheduled surgery during the study (except for bile duct drainage)
3. Ascites of moderate, severe, or requiring drainage
4. Proteinuria of ≥ 2+ on dipstick testing (Grade ≤ 1 confirmed by quantitative assessment is eligible)
5. Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of study drug
6. New York Heart Association congestive heart failure of class II or above, unstable angina, myocardial infarction, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months from the first dose of study drug
7. A prolonged QT/QTc interval (QTcF > 480 ms)
8. Known to be human immunodeficiency virus (HIV) positive
9. Active infection requiring systemic treatment
10. Bleeding or thrombotic disorders or chronic systemic use of anticoagulants requiring therapeutic INR monitoring, eg, warfarin or similar agents (treatment with low molecular weight heparin is permitted)
11. Gastrointestinal bleeding event or active hemoptysis (bright red blood of at least 0.5 teaspoon) within 21 days prior to the first dose of study drug
12. Active malignancy (except for BTC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, carcinoma in-situ of the cervix, or early stage gastric/colorectal cancer) within the past 24 months prior to the first dose of study drug
13. Diagnosed with meningeal carcinomatosis
14. Participants with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 28 days prior to the first dose of study drug. Any signs (eg, radiologic) or symptoms of brain metastases must be stable for at least 28 days prior to the first dose of study drug.
15. Known intolerance to the study drug or any of the excipients
16. History of drug or alcohol dependency or abuse within the last 24 months prior to the first dose of study drug
17. Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study
18. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive human chorionic gonadotropin [hCG or B-hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 3 days before the first dose of study drug.
19. For either males unless undergoing a successful vasectomy (confirmed azoospermia) or females of childbearing potential, the participant and his/her partner do not agree to use a medically appropriate method of contraception throughout the entire study period

    * the use of condom, contraceptive sponge, contraceptive foam, contraceptive jelly, diaphragm, or intrauterine device, otherwise using oral contraceptive (percutaneous or transvaginal also allowed) for at least 28 days before the first dose of study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Yokohama, Kanagawa
  - Ina-machi, Saitama
  - Chuo-ku, Tokyo
  - Koto-ku, Tokyo
  - Mitaka, Tokyo

REFERENCES:
- [Derived] Ueno M, Ikeda M, Sasaki T, Nagashima F, Mizuno N, Shimizu S, Ikezawa H, Hayata N, Nakajima R, Morizane C. Phase 2 study of lenvatinib monotherapy as second-line treatment in unresectable biliary tract cancer: primary analysis results. BMC Cancer. 2020 Nov 16;20(1):1105. doi: 10.1186/s12885-020-07365-4. PMID 33198671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Japan from 23 Oct 2015 to 27 Feb 2019.
Pre-assignment Details: A total of 29 participants were screened and enrolled, of which 3 were screen failures and 26 were treated in the study.
Groups:
- Lenvatinib 24 mg: Participants received lenvatinib 24 milligram (mg) capsules, orally, once daily in 28-days treatment cycles until disease progression, adverse events (AEs), withdrawal of consent, or participant's choice (up to Cycle 40).
Period: Overall Study
Arm/Group | Lenvatinib 24 mg
Started | 29
Treated | 26
Completed | 26
Not Completed | 3
Not completed — Participants did not receive treatment | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included the group of participants who received at least one dose of study drug.
Groups:
- Lenvatinib 24 mg: Participants received lenvatinib 24 mg capsules, orally, once daily in 28-days treatment cycles until disease progression, AEs, withdrawal of consent, or participant's choice (up to Cycle 40).
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. ORR was defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR). Confirmation of CR or PR was performed at least 28 days following the initial achievement of the response.
Time Frame: From the date of first dose of study drug to the date of last documentation of disease progression or date of death from any cause, whichever occurred first (up to approximately 1 year 1 month)
Population: The FAS included the group of participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
percentage of participant | 11.5 [2.4 to 30.2]

2. Secondary Outcome: Progression-free Survival (PFS) Rate at 12 Weeks
Description: PFS was assessed by the investigator based on RECIST 1.1. PFS was defined as the time from the date of first dose to the date of last documentation of disease progression or death from any cause, whichever occurred first. PFS rate was cumulative probability for event-free participants at 12 weeks. PFS rate at 12 weeks was calculated using Kaplan-Meier method.
Time Frame: From the date of first dose to the date of last documentation of disease progression or death from any cause, whichever occurred first (up to Week 12)
Population: The FAS included the group of participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
percentage of participant | 72.2 [50.4 to 85.7]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was assessed by the investigator based on RECIST 1.1. PFS was defined as the time from the date of first dose to the date of last documentation of disease progression or date of death from any cause, whichever occurred first. For participants who did not have an event, PFS were censored. PFS was calculated using Kaplan-Meier method.
Time Frame: From the date of first dose of study drug to the date of last documentation of disease progression or date of death from any cause, whichever occurred first (up to approximately 3 years 4 months)
Population: The FAS included the group of participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
months | 3.19 [2.79 to 7.23]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death from any cause. For the participants who were alive or unknown, OS was censored on the last date participant was known to be event-free or date of data-cut-off. OS was calculated using the Kaplan-Meier method.
Time Frame: From the date of first dose of study drug to the date of death from any cause (up to approximately 3 years 4 months)
Population: The FAS included the group of participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
months | 7.35 [4.50 to 11.27]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was assessed by the investigator based on RECIST 1.1. DCR was defined as the percentage of participants whose BOR was CR, PR or SD.
Time Frame: as for outcome 3
Population: The FAS included the group of participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
percentage of participant | 84.6 [65.1 to 95.6]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was assessed by the investigator based on RECIST 1.1.CBR was defined as percentage of participants with BOR of CR, PR or durable SD. Durable SD: Durable SD: duration of SD greater than or equal to (>=23) weeks.
Time Frame: From the date of first dose of study drug to the date of the last documentation of disease progression or death from any cause, whichever occurred first (up to approximately 3 years 4 months)
Population: The FAS included the group of participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
percentage of participant | 38.5 [20.2 to 59.4]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From signing of informed consent form to 30 days after the decision to discontinue study treatment or 30 days after last dose of study drug, whichever comes later (up to approximately 3 years 4 months)
Population: The safety analysis set included group of participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
participants
  TEAEs | 26
  SAEs | 18

8. Secondary Outcome: Plasma Concentrations of Lenvatinib
Time Frame: Cycle 1 Day 1: 0.5-2 hours post dose (Cycle length is 28 days)
Population: The safety analysis set included group of participants who received at least one dose of study drug. The safety analysis set was used for plasma lenvatinib concentration calculation.
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 26
nanogram per milliliter (ng/mL) | 3.90 [NA to 782] — The lower limit value was not estimable as it was below the limit of quantification.

ADVERSE EVENTS:
Time Frame: From signing of informed consent form to 30 days after the decision to discontinue study treatment or 30 days after last dose of study drug, whichever comes later (up to approximately 3 years 4 months)
Arm/Group | Lenvatinib 24 mg
All-Cause Mortality (participants affected / at risk) | 17/26
Serious Adverse Events (participants affected / at risk) | 18/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 24 mg (N=26)
Abdominal distension (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 2
Bile duct stenosis (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 4
Cholecystitis 1 (Hepatobiliary disorders) | 1
Haemobilia (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Biliary tract infection (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Completed suicide (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal impairment 1 (Renal and urinary disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 24 mg (N=26)
Anaemia (Blood and lymphatic system disorders) | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Hypoparathyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 12
Conjunctival haemorrhage 1 (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 4
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 1
Fistula of small intestine (Gastrointestinal disorders) | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis 4 (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Catheter site pain (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 13
Malaise (General disorders) | 5
Medical device pain (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 8
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 2
Angular cheilitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 2
Lung abscess (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Blood thyroid stimulating hormone increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Thyroxine free increased (Investigations) | 1
Tri-iodothyronine free increased (Investigations) | 1
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 14
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Akathisia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Muscle spasticity (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 16
Renal impairment (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 22
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No